CLINICAL TRIAL: NCT06153719
Title: The Effects of a 12-week Combined Exercise Intervention on the Gut Microbiome of Older Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nottingham Trent University (Other)
Collaborators: University of Reading (Other)
Responsible Party: Principal Investigator, Catarina Ramos, Academic Associate, Nottingham Trent University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1772160
Record Dates: First submitted 2023-11-22; First posted 2023-12-01 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Physical Inactivity
Keywords: Gut microbiome; Exercise; Physical activity; Physical inactivity; Older adults; Gut microbiota
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Active Comparator)
  Interventions: Other: 12-weeks combined exercise intervention
- Control group (Placebo Comparator)
  Interventions: Other: 12-weeks combined exercise intervention

INTERVENTIONS:
Other: 12-weeks combined exercise intervention — This 12-week combined exercise intervention will consist of 3 supervised exercise classes per week, each one lasting 50 minutes. It will involve both aerobic and resistance training in order to follow the UK's physical activity recommendations

SUMMARY:
There are trillions of microorganisms living alongside us in our guts. Recent research has shown that this community, known as the gut microbiome, has a big influence on our health and wellbeing. Imbalances in the composition of the gut microbial community has been linked to several diseases including COVID, mental ill health, and diabetes. When the composition of the gut microbiome changes towards a less healthy one (called dysbiosis) this will, in turn, affect our health in a negative way. The composition of our gut microbiome remains fairly stable during adulthood, however, as we move into older age, there is a shift and its composition will change to a less healthy one; this is one of the reasons why older people can be more susceptible to diseases. Fortunately, there are several tools that we can use to improve our gut microbiome and one of them is exercise. Besides its well-known effects on our health, exercise has been shown to be able to improve the gut microbiome composition of younger people and those with certain metabolic diseases such as obesity. However, less is known about the effects of exercise on the gut microbiome of older adults. The aim of this study, therefore, is to assess the effects of a 12-week exercise intervention on the gut microbiome of physically inactive older adults. Hopefully, after this study, the investigators will have more information on whether exercise can be used as a tool to improve the gut microbiome of older adults therefore improving their overall health and quality of life.

DETAILED DESCRIPTION:
The gastrointestinal (GI) tract, as well as the microbes that live and thrive there, were once thought to be just part of an organ whose only function was food digestion. However, during the last decade, increasing evidence demonstrates that the microbes that reside in the GI tract do a lot more than just digesting food. They have the ability to shape numerous host physiological systems, such as immune function, and to contribute to a healthy ageing process. Moreover, they may be involved in the pathophysiology of several diseases of both acute (e.g., acute respiratory infection, food poisoning) and chronic (e.g., inflammatory bowel disease, asthma, depression, metabolic disease) nature. Key to this influence on host health are the composition and functional activity of the gut microbial community. Both of these characteristics are affected by factors such as age, diet, stress, and medication. Thus, the gut microbiome is modifiable, with the potential to impact many aspects of health and wellbeing, both beneficially and detrimentally.

Gut microbiota diversity and composition changes throughout the lifespan. Initial colonization starts at birth and evolves throughout the life of the host, reaching its early stage maturation around 2-3 years old and then remaining relatively stable during adulthood. As the host starts ageing, the gut microbiota composition and activity changes. An ageing gut microbiota is characterized by a reduced diversity, reduced resilience, and large interindividual variability. Of specific interest to host health is the reduced abundance of Bifidobacteria and Lactobaccilli, and an increased abundance of pathobionts. These changes result in an imbalanced gut microbiota composition - called dysbiosis - and is associated with unhealthy ageing.

There are several factors that may contribute to dysbiosis in older age, such as changes in taste sensation, a decrease in saliva production and weakened chewing strength that altogether may lead to consumption of a more monotonous diet. This, combined with reduced appetite and thus reduced nutrient and energy intake (phenomena called "anorexia of aging"), alterations in the gut physiology (reduced intestinal motility), the presence of antibiotic treatments, consumption of NSAIDs, polypharmacy, a weakened immune system and living arrangements will ultimately lead to an imbalanced microbiota, thus resulting in dysbiosis.

In a dysbiotic gut, a number of microbial mediated changes can impact on the health of the host. For example, pathogenic bacteria can disturb the intestinal barrier, and their sub-products, such as bacterial lipopolysaccharide (LPS) can enter the systemic circulation and cause chronic inflammation. This, combined with the persistent chronic low grade inflammation that occurs with age (known as 'inflammaging') and the immunosenescence that occurs during the ageing process, will increase the inflammatory state and can contribute to several diseases/conditions, such as obesity, diabetes type 1, diabetes type 2, inflammatory bowel diseases (IBD), frailty, insulin resistance, cardiovascular diseases (CVDs), asthma, colorectal cancer, stress-related disorders, dementia, hypertension, Alzheimer's disease, Parkinson's disease and rheumatoid arthritis. Furthermore, perturbations in this tightly regulated ecosystem will affect energy metabolism, nutrient absorption, appetite regulation, the immune system, and the synthesis of several key metabolites, such as short chain fatty acids (SCFAs) and vitamins. Therefore, interventions to change the gut microbiome to a 'younger', less dysbiotic profile are desirable in older adults as part of successful aging.

In the current project, which forms part of a Doctoral research programme, we are interested in whether exercise/physical activity (PA) can positively influence the composition and functional activity of the gut microbiome of older adults. Although a relatively new area of research, several studies have shown that PA and exercise are associated with an altered gut microbiome both in terms of microbial composition and functional activity in younger populations. For example, a study compared the gut microbiota composition of professional rugby athletes with sedentary controls and verified that their microbiotas were distinctly different. Athletes had higher microbial diversity, higher SCFA producing bacteria and an increased abundance of health-related pathways when compared to the sedentary controls. The same conclusion was reached by another research group who found that pre-menopausal women who were active had a different microbiota composition when compared to women who were sedentary. More specifically, healthy women had a higher abundance of health-promoting bacterial species, such as Faecalibacterium prausnitzi, Roseburia hominis and Akkermansia muciniphila. Moreover, they also found an inverse association between microbial diversity and sedentary behaviour and a correlation between body fat, age, muscle mass and physical activity with several bacterial populations. These previous studies demonstrate that physical activity is associated with a health-associated gut microbiota, however, none of them controlled for the influence of diet as a confounding factor. In fact, it is possible that people who are physically active tend to have a healthier diet when compared to inactive or sedentary people, and this can affect the results. A research group, however, demonstrated that 6 weeks of endurance exercise training was able to induce changes in the gut microbiota in lean but not in obese subjects independently of the diet, suggesting that exercise/PA can indeed induce changes in the gut microbiome composition per se. In the previous study, exercise was able to increase the concentration of SCFAs and the bacteria that produce them. However, the exercise-induced changes in the gut microbiota returned to baseline after a 6-week washout period, during when the participants' returned to their sedentary lifestyle. These findings suggest that the sustainment of exercise may be needed in order to maintain, or improve, the beneficial changes that occur in the gut microbiota.

Focusing now on studies performed in older adults, little is known about the effects of exercise/PA or sedentary behaviour on the gut microbiome with only 9 publications so far, consisting of 3 intervention studies, two performed in Asia and one in the USA and 6 observational studies, performed in Sweden, USA, Israel, Ireland and Slovakia. A recently published systematic review of the effects of exercise and PA on the gut microbiome of older adults produced by our research group which aimed to summarise the results of humans studies performed in this topic, found that exercise/PA was able to increase the abundance of health related bacteria and decrease the abundance of harmful bacteria, and that older people who were more active tended to have a better gut microbiota composition containing more health-related bacteria than when compared with their inactive counterparts. However, due to methodological disparities between studies, it was hard to find a consensus on which taxa were most responsive to/associated with PA/exercise. Based on the information gathered on that systematic review, some recommendations were made regarding future studies in the field, such as the need to perform more observational studies in western populations (since the majority of publications are in Asian populations), the need to perform high quality exercise intervention studies by controlling some important confounding factors (such as diet and body composition) in older adults and by including different types of exercise. Another avenue would be to assess the effects of sedentary behaviour on the gut microbiome of older adults, since it has been previously shown that inactive people have a different gut microbiome composition when compared to their active counterparts.

Our research group is currently conducting an observational study which aims to compare the gut microbiome composition of physically active vs physically inactive community dwelling older adults. We want to investigate if exercise/PA has a beneficial effect on the gut microbiome of a sample of 100 UK older adults and assess if there is any association between body composition, cardiorespiratory fitness, and physical function with certain bacterial taxa.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 65-85 years old
* Healthy, free-living individuals
* Vaccinated against COVID-19
* Physically inactive (<150 mins/week of PA)
* No participation in any exercise intervention studies in the last 3 months
* BMI Between 20-35 kg/m2

Exclusion Criteria:

* The use of antibiotics 3 months before or during the study
* Cancer
* Intestinal inflammatory conditions (e.g., Crohns, ulcerative colitis)
* Consumption of proton pump inhibitors (e.g., omeprazole, lansoprazole, etc…)
* Auto-immune diseases
* GI diseases (e.g., IBS, peptic ulcers)
* Routine consumption of pre and/or probiotic foods or supplements
* On blood thinners

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Gut microbiome composition | At the begining and at the end of the intervention
  Gut microbiome composition will be analysed using 16s rRNA sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Kirsty Hunter, Principal Investigator — Nottingham Trent University
Locations (1):
- Nottingham Trent University - Clifton campus, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ramos C, Gibson GR, Walton GE, Magistro D, Kinnear W, Hunter K. Systematic Review of the Effects of Exercise and Physical Activity on the Gut Microbiome of Older Adults. Nutrients. 2022 Feb 5;14(3):674. doi: 10.3390/nu14030674. PMID 35277033
- [Background] Taniguchi H, Tanisawa K, Sun X, Kubo T, Hoshino Y, Hosokawa M, Takeyama H, Higuchi M. Effects of short-term endurance exercise on gut microbiota in elderly men. Physiol Rep. 2018 Dec;6(23):e13935. doi: 10.14814/phy2.13935. PMID 30536648
- [Background] Erlandson KM, Liu J, Johnson R, Dillon S, Jankowski CM, Kroehl M, Robertson CE, Frank DN, Tuncil Y, Higgins J, Hamaker B, Wilson CC. An exercise intervention alters stool microbiota and metabolites among older, sedentary adults. Ther Adv Infect Dis. 2021 Jun 25;8:20499361211027067. doi: 10.1177/20499361211027067. eCollection 2021 Jan-Dec. PMID 34262758
- [Background] Barton W, Penney NC, Cronin O, Garcia-Perez I, Molloy MG, Holmes E, Shanahan F, Cotter PD, O'Sullivan O. The microbiome of professional athletes differs from that of more sedentary subjects in composition and particularly at the functional metabolic level. Gut. 2018 Apr;67(4):625-633. doi: 10.1136/gutjnl-2016-313627. Epub 2017 Mar 30. PMID 28360096
- [Background] Bressa C, Bailen-Andrino M, Perez-Santiago J, Gonzalez-Soltero R, Perez M, Montalvo-Lominchar MG, Mate-Munoz JL, Dominguez R, Moreno D, Larrosa M. Differences in gut microbiota profile between women with active lifestyle and sedentary women. PLoS One. 2017 Feb 10;12(2):e0171352. doi: 10.1371/journal.pone.0171352. eCollection 2017. PMID 28187199
- [Background] Allen JM, Mailing LJ, Niemiro GM, Moore R, Cook MD, White BA, Holscher HD, Woods JA. Exercise Alters Gut Microbiota Composition and Function in Lean and Obese Humans. Med Sci Sports Exerc. 2018 Apr;50(4):747-757. doi: 10.1249/MSS.0000000000001495. PMID 29166320